CLINICAL TRIAL: NCT01622322
Title: Effect Nitrous Oxide On Acute Postoperative Pain and Opioid Consumption and Chronic Pain After Inguinal Hernia Repair Surgery
Brief Title: Nitrous Oxide On Acute Postoperative Pain and Opioid Consumption and Chronic Pain After Inguinal Hernia Repair Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no enrollment
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Alparslan Turan, PI, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 10/1539
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Inguinal Hernia Repair; Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Nitrous Oxide; Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitrous oxide (Experimental): Subjects will receive General anesthesia with Nitrous Oxide.
  Interventions: Drug: Nitrous Oxide
- Oxygen (Placebo Comparator): Subjects will receive General anesthesia with oxygen.
  Interventions: Other: oxygen

INTERVENTIONS:
Drug: Nitrous Oxide — Nitrous Oxide, 70%, O2 30%) 1-5 L, Sevoflurane 1-2%, ETCO2: 32-35 mmHg.
  Arms: Nitrous oxide
Other: oxygen — Subjects will receive General anesthesia: (Air, 70%, O2 30%) 1-5 L, Sevoflurane 1-2%, ETCO2: 32-35 mmHg.
  Arms: Oxygen

SUMMARY:
To compare postoperative pain, opioid consumption and chronic pain in patients undergoing to hernia repair surgery after receiving nitrous oxide or oxygen during the general anesthesia.

DETAILED DESCRIPTION:
The study is prospective and double blind. In the clinic, patients undergoing inguinal hernia surgery that meet the criteria for inclusion into the study and agreed to participate in the study will be randomized into two groups. In the first group of patients will receive Nitrous Oxide and In the second group of patients will receive oxygen during the general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old at time of the first procedure
* American Society of Anesthesiologists physical status I or II
* Inguinal hernia repair surgery undergoing the general anesthesia

Exclusion Criteria:

* Neuropathic disease
* Chronic opioid users
* Contraindication for Nitrous Oxide receive
* Consent will not be obtained patient
* Psychiatric disorders
* Current or recent drug abuse (within past 6 months).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Nitrous oxide and chronic pain | 30 days post operative
  The effect of 70% N20/30% O2 on post inguinal hernia repair procedure in prevention of chronic pain.
Nitrous oxide and opioid consumption | 4 hours after surgery
  The effect of 70% N20/30% O2 on post inguinal hernia repair procedure in decrease in opioid consumption.

SECONDARY OUTCOMES:
smoking and post operative pain | 4 hours after surgery
  The effect of active smoking to increase post operative acute pain.
smoking and chronic pain | 30 days post operative
  The effect of active smoking and chronic pain

CONTACTS AND LOCATIONS:
Overall Officials: Alparslan Turan, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Gulhane Military Medical Academy Hospital, Etlik, Ankara, Turkey (Türkiye)